CLINICAL TRIAL: NCT06771115
Title: A Phase 2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VTX3232 Alone or in Combination With Semaglutide in Participants With Obesity
Brief Title: Phase 2a Placebo-Controlled Study of VTX3232 Alone or in Combination With Semaglutide in Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zomagen Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VTX3232-204
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Obesity
Keywords: NLRP3 Inhibitor; VTX3232; Zomagen
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will employ a double-blind design for study treatment tablets (i.e., VTX3232 or Placebo); assignment to treatment group with semaglutide injections plus study treatment tablets or to treatment group with study treatment tablets alone will not be blinded. Participants, Investigators, study center staff, persons performing the assessments, and the Sponsor are to remain blinded to the identity of the study treatment tablets from the time of randomization until the database lock for the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VTX3232 Dose A (Experimental): VTX3232 Dose A
  Interventions: Drug: VTX3232 Dose A
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- VTX3232 Dose A in combination with semaglutide (Experimental): VTX3232 Dose A in combination with semaglutide
  Interventions: Drug: VTX3232 Dose A in combination with semaglutide
- Placebo in combination with semaglutide (Experimental): Placebo in combination with semaglutide
  Interventions: Drug: Placebo in combination with semaglutide

INTERVENTIONS:
Drug: VTX3232 Dose A — VTX3232 Dose A
  Arms: VTX3232 Dose A
Drug: Placebo — Placebo
  Arms: Placebo
Drug: VTX3232 Dose A in combination with semaglutide — VTX3232 Dose A in combination with semaglutide
  Arms: VTX3232 Dose A in combination with semaglutide
Drug: Placebo in combination with semaglutide — Placebo in combination with semaglutide
  Arms: Placebo in combination with semaglutide

SUMMARY:
This is a study to understand if taking VTX3232 alone or in combination with semaglutide is safe in participants diagnosed with Obesity. Approximately 160 patients will take VTX3232 Dose A, Placebo, VTX3232 Dose A in combination with semaglutide, or Placebo in combination with semaglutide.

This study consists of a 30-day Screening Period (to see if a participant qualifies for a study), a 12-week double-blind treatment period (a participant receives VTX3232 Dose A, Placebo, VTX3232 Dose A in combination with semaglutide, or Placebo in combination with semaglutide), and a 30-day Follow-Up Period. The maximum duration of treatment will be approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants are male or female ≥ 18 years up to ≤ 80 years of age.
* Ability to comply with study requirements.
* BMI ≥ 30.0 to ≤ 42.0 kg/m2 at screening.
* Stable body weight (± 5%) for at least 3 months prior to screening.
* hs-CRP ≥ 2 mg/L at screening.
* Hypertension or hyperlipidemia which are known to be associated with increased risk of cardiovascular events, if present, must be controlled with stable dose/therapy.
* History of at least one self-reported unsuccessful dietary effort to lose body weight.

Exclusion Criteria:

* Obesity induced by endocrinologic disorders, or diagnosed genetic or syndromic forms of obesity
* Have any prior diagnosis of diabetes mellitus
* Current participation (or within the last 3 months) in an organized weight reduction program.
* History or presence of clinically significant gastric emptying abnormality (e.g., severe gastroparesis or gastric outlet obstruction) or chronically take drugs that directly affect GI motility, have undergone prior surgical treatment for obesity (e.g., gastric bypass [bariatric] surgery or restrictive bariatric surgery), or have an endoscopic and/or device-based therapy for obesity.
* Clinically relevant medical condition(s) that put the participant at risk or will make implementation of the protocol or interpretation of the study difficult.
* Use of any medication (e.g., GLP-1 agonists), nutritional supplement, or over the counter product for weight loss within the previous 6 months or during study participation, unless administered as a part of assigned study treatment in this study.
* Receipt of the following medications:

  1. Any immunosuppressive biologic or targeted therapy within 90 days prior to Day 1.
  2. Use of anti-inflammatory medications within 30 days prior to Day 1
  3. Colchicine within 30 days prior to Day 1.
  4. Glucose-lowering agent(s) administered for conditions other than diabetes within 90 days before screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Incidence Rate and Severity of Adverse Event (AE), Serious Adverse Event (SAE), and AEs leading to study treatment discontinuation through study completion | Day 1 of treatment period through study completion, up to 16 weeks
  Incidence of AEs and SAEs and AEs leading to study treatment discontinuation

SECONDARY OUTCOMES:
Change from baseline in hs-CRP level | Day 1 of treatment period to week 12 of treatment period
  Change from baseline in hs-CRP through 12 weeks of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Naik, PhD, Study Director — Zomagen Biosciences Ltd.
Locations (14):
- United States (14):
  - 840005, Birmingham, Alabama
  - 840003, Lake Forest, California
  - 840011, Long Beach, California
  - 840001, Largo, Florida
  - 840012, Ocoee, Florida
  - 840016, Port Orange, Florida
  - 840014, Newton, Kansas
  - 840015, Marrero, Louisiana
  - 840017, Marrero, Louisiana
  - 840002, Austin, Texas
  - 840006, Dallas, Texas
  - 840013, San Antonio, Texas
  - 840018, San Antonio, Texas
  - 840010, Waco, Texas

IPD SHARING:
Plan to Share IPD: Undecided